CLINICAL TRIAL: NCT05984368
Title: First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation and Multiple Dose Escalation Phase I Clinical Trial of BG136 for Injection in Healthy Subjects
Brief Title: A Clinical Study of BG136 Injection in Healthy Chinese Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of Clinical Trials Center of Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG136211213
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single-dose and multi-dose, dose escalation, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): A single ascending dose (SAD) study divided into 7 dose groups: 2 mg (exploratory dose), 24 mg, 50 mg, 100 mg, 200 mg, and 300 mg, 400 mg (optional dose group), with 2 mg enrolling 2 subjects (all receiving the test drug) and the remaining 8 subjects in each group (6 test drug, 2 placebo).
  Interventions: Drug: BG136; Drug: Placebo
- Part 2 (Experimental): Multiple ascending dose (MAD) study, divided into 3 dose groups: 100 mg, 200 mg and 300 mg, each group included 8 healthy subjects (6 test drug, 2 placebo).
  Interventions: Drug: BG136; Drug: Placebo

INTERVENTIONS:
Drug: BG136 — Subjects injected with BG136 in Part 1 and Part 2
Drug: Placebo — Subjects injected with Placebo in Part 1 and Part 2

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled trial in healthy subjects. The trial consisted of two parts: part 1: single ascending dose (SAD) study and part 2: multiple ascending dose (MAD) study. Each part had multiple Intravenous infusion administration dose groups. Prior to the formal initiation of the dose-escalation trial, the safety, tolerability, and pharmacokinetics (PK) characteristics of a pretest dose (pilot dose) of 2 mg will be evaluated in 2 subjects (both administered BG136 for injection)

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blind, placebo-controlled clinical trial in healthy subjects. The trial consists of two parts: Part 1: a single ascending dose (SAD) study with seven dose groups: 2 mg (exploratory dose), 24 mg, 50 mg, 100 mg, 200 mg, and 300 mg, 400 mg (optional dose groups), with two subjects enrolled in the 2 mg group (all receiving the test drug), and eight subjects enrolled in each of the remaining groups (six test drug and two placebo); Part 2: a multiple ascending dose (MAD) study with seven dose groups: two subjects (six test drug and two placebo); and Part III: a randomized, double-blind, placebo-controlled clinical trial in healthy subjects, with a randomized, double-blind, placebo-controlled clinical trial in healthy subjects. Part II: Multiple ascending dose (MAD) study, divided into 3 dose groups: 100 mg, 200 mg and 300 mg, each including 8 healthy subjects (6 test drug, 2 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female subjects aged 18-55 years (including the threshold);
* Weight ≥ 50 kg for men and ≥ 45 kg for women and body mass index (BMI): 19.0-26.0 kg/m2 (including borderline values);
* Subjects understand and comply with the study process, can communicate well with the investigator, volunteer to participate in the trial and sign an informed consent form.

Exclusion Criteria:

* Diseases to be excluded due to clinical abnormalities within 3 months prior to screening, including but not limited to neurological/psychiatric, cardiovascular, hematological and lymphatic, immune, gastrointestinal, urinary, endocrine, metabolic, and skeletal conditions. History of diseases of the urinary, endocrine, respiratory, metabolic and skeletal systems.
* History of comorbid gastrointestinal related disorders
* Those who have had surgery within 3 months prior to screening or plan to have surgery during the study period；
* Screening subjects whose vital signs, physical examination, routine blood, urine, blood biochemistry, coagulation function, and electrocardiogram are judged by the investigator to be abnormal and clinically significant；
* Subject's imaging determined by the investigator to be clinically significant for abnormalities；
* Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody screening, human immunodeficiency virus (HIV) antibody screening, treponema pallidum antibody (TP-Ab) any test positive；
* History of food or drug allergies or other allergic diseases；
* History of substance abuse in the 12 months prior to screening, or drug use in the 3 months prior to screening, or a positive urine drug screen；
* Positive breath test results for alcohol or regular alcohol consumption in the 6 months prior to screening, i.e., an average of more than 14 units of alcohol per week (1 unit ≈ 200 mL of beer at 5% alcohol or 25 mL of spirits at 40% alcohol or 85 mL of wine at 12% alcohol), or inability to abstain from alcohol consumption for 48 hours prior to the first dose of the medication and for the entire study period；
* Smokers who smoked an average of ≥5 cigarettes per day in the 3 months prior to screening or who could not give up smoking 48 hours prior to the first dose and throughout the study period；
* Those who have received a blood transfusion or used blood products ≥ 400 mL or 2 units within 3 months prior to screening, or those who have lost ≥ 400 mL of blood within 6 months, or those who have donated blood within 3 months；
* Participated in another clinical trial within 3 months prior to screening and took the trial drug or used the trial device；
* Any prescription (including vaccines), over-the-counter medications used within 4 weeks prior to screening；
* Those who have used herbal medicines or health supplements for the treatment and/or prevention of their own disease within 2 weeks prior to screening；
* Persons with special dietary requirements who are unable to follow a standardized diet or who are unable to avoid xanthine-rich beverages or foods or fruits or fruit juices that may interfere with metabolism for 48 hours prior to dosing and up to study completion;
* Those who have difficulty in collecting blood from veins or who suffer from needle;
* Women who are pregnant, breastfeeding, or who have had unprotected sex within 2 weeks prior to screening, or who have had a positive pre-test pregnancy test;
* Male subjects (or their partners) or female subjects who are planning a pregnancy, sperm donation, or oocyte donation from the time of signing the Informed Consent Form until 3 months after the end of the administration of the medication;
* Those who do not wish to use one of the medically approved non-pharmacological contraceptives (e.g., intrauterine device or condom) during the trial period;
* Subjects deemed unsuitable by the investigator to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 14 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Peak Plasma Concentration (Cmax) | up to 14 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | up to 14 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | up to 14 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No